CLINICAL TRIAL: NCT06860347
Title: Biomarkers for Fatigue in Patients with Myasthenia Gravis
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Martijn R. Tannemaat, MD PhD, MD PhD, Leiden University Medical Center
Other Study IDs: NL72266.058.20
Record Dates: First submitted 2022-08-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and muscle biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Rationale: Myasthenia Gravis (MG) is a chronic autoimmune disease affecting the neuromuscular junction. Although a hallmark of MG is muscle fatigability due to dysfunction of the neuromuscular junction (peripheral fatigue), a large number of MG patients also report symptoms of central or cognitive fatigue. Central fatigue is defined as an experienced lack of energy, physically and/or mentally. In October 2019 we performed a cross-sectional survey study (P15.287) among 420 Dutch MG patients showing a clinically relevant central fatigue rate of 62% on the Checklist Individual Strength-Fatigue subscale (CIS-f). In this prior study, we identified a number of factors associated with fatigue, but these factors cannot fully explain the observed high prevalence of fatigue in MG and very little is known on its biological substrates and pathophysiology.

Objectives: The main objective is to investigate if there are biomarkers for fatigue in MG. The secondary objective is to investigate the muscle origin of these biomarkers.

Study design: This study will be an exploratory study, subdivided in part I and part II (optional).

Study population: Patients with Myasthenia Gravis recruited after previous participation in the cross-sectional fatigue survey study (P15.287).

Intervention:

Phase I:

Visit 1, time: 0

* blood withdrawal
* muscle biopsy (not mandatory for participation)
* QMG
* questionnaires on medication, disease severity, fatigue, depressive symptoms and physical condition

Phase II (optional):

Visit 2, time: 6-12 months after visit 1, after analysis of phase I results.

* blood withdrawal (similar analysis as phase I)
* QMG
* questionnaires on medication, disease severity, fatigue, depressive symptoms and physical condition

ELIGIBILITY:
Inclusion Criteria:

* Male of female patients aged ≥ 18 years
* Subjects must understand the requirements of the study and provide written informed consent.
* Diagnosis of MG:

  * Clinical signs or symptoms characteristic for MG and
  * A positive serologic test for AChR antibodies

Exclusion Criteria:

A medical history of other active auto-immune disorders for which the patient currently receives a medical treatment, such as thyroid disease or rheumatoid arthritis.

* A medical history of neoplasms within the last year.
* Substance abuse.

Exclusion criteria for muscle biopsy

* The use of anticoagulants therapy.
* Allergy for lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myasthenia Gravis recruited after previous participation in the cross-sectional fatigue survey study (P15.287).
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
blood biomarker | 2022
  To investigate whether there is a potential biomarker, which corresponds with fatigue in MG, among the biomarkers that were previously identified in other disorders. For this objective we aim to determine and compare the diagnostic yield of several serum biomarkers which were (possibly) associated with central fatigue in other disorders in previous studies.

SECONDARY OUTCOMES:
Brain muscle axis | 2022-2023
  To investigate whether a potential biomarker, which corresponds with fatigue in MG, is derived from muscle tissue. Therefore, we will assess the expressed mRNA in skeletal muscle tissue to confirm the muscle origin of elevated circulating serum biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Tannemaat, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruiter AM, Verschuuren JJGM, Tannemaat MR. Prevalence and associated factors of fatigue in autoimmune myasthenia gravis. Neuromuscul Disord. 2021 Jul;31(7):612-621. doi: 10.1016/j.nmd.2021.04.002. Epub 2021 Apr 24. PMID 34034925
- [Background] Ruiter AM, Verschuuren JJGM, Tannemaat MR. Fatigue in patients with myasthenia gravis. A systematic review of the literature. Neuromuscul Disord. 2020 Aug;30(8):631-639. doi: 10.1016/j.nmd.2020.06.010. Epub 2020 Jul 1. PMID 32718868